CLINICAL TRIAL: NCT06553846
Title: A Clinical Trial on Pharmacokinetics and Radiation Dosimetry, Safety and Preliminary Efficacy Evaluation of Lutetium [177Lu]-FAP-75 for the Treatment of Patients With Advanced Solid Tumors
Brief Title: A Clinial Trial of Lutetium [177Lu]-FAP-75 for the Treatment of Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [177Lu]-FAP-75-001
Record Dates: First submitted 2024-08-02; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumors
Keywords: solid tumors; FAP; Radionuclide therapy
MeSH Terms: interventions — Lutetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Lutetium [177Lu]-FAP-75 accumulates at the tumor site, and beta rays act on surrounding tumor cells, causing tumor cell apoptosis.
  Interventions: Drug: Lutetium [177Lu]-FAP-75

INTERVENTIONS:
Drug: Lutetium [177Lu]-FAP-75 — Lutetium [177Lu]-FAP-75 will be administrated per dose level in which the patients are assigned.

SUMMARY:
To explore the safety, tolerability, initial efficacy, pharmacokinetic profile and radiation dosimetry of lutetium [177Lu]-FAP-75 in the treatment of patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a prospective, open, dose-exploring clinical study of Lutetium [177Lu]-FAP-75 in the treatment of patients with advanced solid tumors. The study was divided into two stages, the first stage was dose exploration study, and the second stage was case expansion study. In the first phase of this study, several dose groups were designed. Subjects may receive only one of these doses and may not receive multiple doses in the same subject. The drug was administered every 6 weeks, and the DLT observation period was 6 weeks after the first dose. Firstly, the first dose safety introduction of human body was carried out. Based on the results of the preclinical study of this product, an appropriate number of enrolled subjects in the first and second stages were selected to enter the PK and radiation dosimetry detection groups. After the end of the DLT observation period, subjects who met the criteria for continued dosing were allowed to continue to receive the investigational drug therapy for subsequent cycles. For all participants enrolled in this study, the study process included a screening period, a treatment period and a follow-up period. In the course of the trial, extended studies of other tumor species can be conducted based on new advances and results of clinical studies of similar drugs to further explore the safety, tolerability and initial effectiveness of specific tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical trial, understand the research procedure and be able to sign the informed consent in person;
2. Age 18-80 years old (including 18 and 80 years old), gender is not limited;
3. ECOG score 0-1;
4. The expected survival period is not less than 4 months;
5. Subjects with solid tumors diagnosed histologically or cytologically at advanced stage (unresectable or metastatic) after failure of standard treatment (disease progression or intolerance) or lack of effective treatment are enrolled in this study.
6. There must be at least one measurable target lesion (according to RECIST V1.1);
7. Positive lesion uptake in FAP PET/CT imaging
8. The level of vital organ function meets the following requirements :

   * Neutrophil ≥1.5×109/L;
   * Platelets ≥100×109/L;
   * Hemoglobin ≥90g/L;
   * Total bilirubin ≤1.5×ULN; If there is biliary obstruction or Gilbert syndrome, total bilirubin ≤3×ULN;
   * ALT and AST≤3 x ULN; If liver metastasis exists, ALT and AST≤5×ULN;
   * Serum albumin ≥30g/L;
   * Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 ml/min (calculated according to Cockcroft-Gault formula);
   * INR≤1.5×ULN and APTT≤1.5×ULN (for subjects not receiving anticoagulant therapy, stable therapy dose is required for subjects receiving anticoagulant therapy).
9. Women of childbearing age must undergo a blood pregnancy test within 72 hours before the first dosing, must be non-lactating.

Exclusion Criteria:

1. Known significant weight loss (>10%) within 28 days prior to signing the informed consent.
2. Prior and follow-up treatment:

   1. Received any radionuclide therapy or radiotherapy within 6 months before enrollment.
   2. Prior treatment with any FAP target nuclide.
   3. Received anti-tumor therapy such as surgery (except diagnostic biopsy and drainage of serosal effusion), chemotherapy, immunotherapy, and monoclonal antibodies within 4 weeks prior to admission; received anti-tumor endocrine drugs within 2 weeks; received nitrosourea or mitomycin chemotherapy within 6 weeks; eluted oral targeted therapy drugs with less than 5 half-lives or 4 weeks (whichever is shorter).
   4. Received any other investigational drug treatment within 4 weeks prior to enrollment.
   5. Any surgical procedures requiring general anesthesia and significant incisions (e.g., central venous access, percutaneous feeding tube insertion) within 6 weeks of enrollment (expected surgery).
3. Combined with the following diseases:

   1. Patients with meningeal metastasis or diffuse central nervous system metastasis or active central nervous system metastasis who require any radiotherapy, gamma knife, surgery, or medication to control the symptoms of metastasis 1 month prior to screening are excluded. Patients with a limited number of stable central nervous system metastases could be enrolled.
   2. severe urinary incontinence, hydronephrosis, and severe urination dysfunction. Note: Subjects with bladder outflow tract obstruction that can be controlled with the best available standard of care are eligible for study participation.
   3. Co-active hepatitis B, hepatitis C.
   4. Known to have acquired immune deficiency syndrome (AIDS) or tested positive for HIV.
   5. Active syphilis infection.
4. Known allergy to components of the investigatory drug or its analogues.
5. Malignancies outside the target tumor species that are expected to alter life expectancy or may interfere with disease assessment within the first 5 years of enrollment. The exception is for cured malignancies with a low risk of metastasis and death, such as non-metastatic skin basal cell carcinoma or skin superficial squamous cell carcinoma.
6. Serious infections occurred within 4 weeks prior to enrollment, such as severe pneumonia requiring hospitalization, bacteremia, infection complications, etc., and signs and symptoms of infection within 2 weeks prior to enrollment requiring intravenous antibiotic treatment (except for prophylactic antibiotic use).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-19 (Estimated); Primary Completion 2025-02-18 (Estimated); Study Completion 2025-08-18 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | Up to approximately 12 months
  Evaluated by RECIST1.1
Adverse events(AEs) | From the first drug administration to within 90 days for the last drugs dose
  AEs , are assessed by NCI-CTCAE v5.0
Dose Limiting Toxicity(DLT) | within 6 weeks from the first drug administration
  Dose Limiting Toxicity are assessed by NCI-CTCAE v5.0
Second-stage dose | through study completion, an average of 1 year
  Second-stage dose is the recommend dose for the second stage of this trial which is determined by the safety profile of the first stage of this trial.

SECONDARY OUTCOMES:
Overall survival(OS) | Up to approximately 12 months
  Time from the date of enrollment to date of death from any cause.
Disease Control Rate(DCR) | Up to approximately 12 months
  Evaluated by RECIST1.1
Duration of Response(DoR) | Up to approximately 12 months
  Evaluated by RECIST1.1
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  PFS is defined as the time from the date of first dose of study drug to the date of the first documentation of disease progression or date of death, whichever occurs first.
Radiation dosimetry | Up to 6 weeks
  Dosimetry, measured as absorbed dose in tumor and normal organs (Gy/GBq), was estimated in the first treatment cycle for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center;Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided